CLINICAL TRIAL: NCT04454775
Title: The Effect of Raloxifene on the Parameters of Coagulation System in the Postmenopausal Women
Brief Title: Raloxifene on Coagulation System in the Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, professor, Karadeniz Technical University
Other Study IDs: 2005/47
Record Dates: First submitted 2020-06-05; First posted 2020-07-01 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Raloxifene; Postmenopausal Women
Keywords: raloxifene; coagulation system; von Willebrand factor; Factor 8; vitamin D; protein C; protein S; antithrombin- III; fibrinogen
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group I: 50 cases who received raloxifene and calcium therapy
  Interventions: Diagnostic Test: coagulation system parameters; factor 8, von Willebrand factor, protein C, protein S, antithrombin III and fibrinogen were studied.
- group II: 30 cases who received only calcium therapy
  Interventions: Diagnostic Test: coagulation system parameters; factor 8, von Willebrand factor, protein C, protein S, antithrombin III and fibrinogen were studied.

INTERVENTIONS:
Diagnostic Test: coagulation system parameters; factor 8, von Willebrand factor, protein C, protein S, antithrombin III and fibrinogen were studied.

SUMMARY:
Objective: The aim of this study is to assess the effects of raloxifene HCl on coagulation parameters in healthy postmenopausal women.

Material and method: 80 healthy postmenopausal women were evaluated at Karadeniz Technical University Hospital at gynecology out-patient clinic from December 2005 to December 2006. Local institutional ethics committee approved our study protocol and written informed consent was obtained from all participants before enrollment. All patients received daily 600 milligrams of calcium and 400 international units of vitamin D (Cal-D-VİTA, Roche Switzerland,). 60 milligrams of raloxifene HCI, which is a selective estrogen receptor modulator (SERM), was added to treatment protocol if patients required hormonal therapy. Patients receiving raloxifene therapy in addition to calcium and vitamin D therapy formed the study group(n=50). Control group (n=30) was made up of the patients only receiving calcium and vitamin D. Factor 8, von Willebrand factor, protein C, protein S, antithrombin- III and fibrinogen levels were measured in all patients before treatment. These measurements were repeated at three and twelve months after treatment. Comparisons were performed with Student t test or Mann Whitney test between the two groups and two-way ANOVA within the groups. Proportions were compared with Fisher exact or Chi-square tests. Statistically analysis was done with SPSS packet program (SPSS 11; SPSS Inc.) All p values were two-tailed and p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* In the study planned on patients who have not had menstruation for at least one year, or who have been in menopause naturally or surgically,
* the presence of menopause was accepted if the patients' FSH level was> 40 IU / L. Verbal and written consent was obtained from all patients included in the study.

Exclusion Criteria:

* . Hypertension,
* diabetes mellitus,
* hypercholesterolemia,
* presence of hepatic-renal-thyroid-parathyroid-adrenal diseases,
* cardiovascular,
* cerebrovascular and thromboembolic diseases,
* undiagnosed vaginal bleeding,
* presence of hormone-dependent malignancy or anamnesis,
* presence of varicose veins,
* chronic drug use that disrupts sex steroid metabolism
* cases with smoking
* alcohol use

Ages: 42 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The treatment of menopause and hormone happens only in female sex.
Study Population: Patients who applied to Menopause outpatient clinic with the approval of Karadeniz Technical University Faculty of Medicine Ethics Committee numbered 2005/47 were evaluated within the scope of the prospective study. Working time was determined as 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2006-12-01 (Actual); Study Completion 2006-12-20 (Actual)

PRIMARY OUTCOMES:
Measuring coagulation parametres | 1 year
  After collecting all blood, Factor 8, von Willebrand factor, protein C, protein S, antithrombin- III, and fibrinogen levels were measured in all patients.